CLINICAL TRIAL: NCT04611425
Title: REmimazolam Infusion in the Context of Hypnotic Shortage in the Critical Care Unit During the Pandemic of COVID-19. The Non-randomized, Non-controlled, Pilot, Open, Mono-centric REHSCU Study
Brief Title: REmimazolam Infusion in the Context of Hypnotic Shortage in the Critical Care Unit During the Pandemic of COVID-19: REHSCU Study
Acronym: REHSCU
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Nantes University Hospital (Other)
Collaborators: Paion UK Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: RC20_0319
Record Dates: First submitted 2020-10-07; First posted 2020-11-02 (Actual); Last update posted 2021-11-04 (Actual); Status verified 2021-10

CONDITIONS: Acute Respiratory Failure; COVID-19; Trauma; Stroke; Sepsis; Shock
Keywords: Remimazolam; Sedation; Shortage; Critical care; COVID-19
MeSH Terms: conditions — COVID-19; Wounds and Injuries; Stroke; Sepsis; Shock | interventions — remimazolam

STUDY DESIGN:
Intervention Model Description: Non-controlled
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Remimazolam (Experimental): Patients will receive an infusion of Remimazolam for a maximum duration of 48 hours.
  The dose of Remimazolam will be adapted according to our ICU protocol of analgesia-sedation management, based on validated scale (Richmond Assessment Sedation Scale)
  Interventions: Drug: Remimazolam

INTERVENTIONS:
Drug: Remimazolam — Patients will receive an infusion of Remimazolam for a maximum duration of 48 hours. The dose of Remimazolam will be adapted according to the ICU units protocol of analgesia-sedation management, based on validated scale (Richmond Assessment Sedation Scale). Owing to previous data gathered through a previous study in Japan, the initial dose of infusion will be within a 0.2-0.5 mg/min range. The dose of Remimazolam can be increased or decreased by 0.1mg/min when needed. The maximum dose of Remimazolam will be set at 1 mg/min.
  Other Names: Remimazolam (CNS 7056)

SUMMARY:
The worldwide COVID-19 pandemic has led to a dramatic increase in the number of patients hospitalized in intensive care units for an acute respiratory failure in all countries. This situation has quickly led to massive shortage in masks, mechanical ventilation machines and common medications such as hypnotics. All countries over the world are currently experiencing a major shortage in basic hypnotic medications (propofol, midazolam) in the intensive care as well as in the operating theatre. The Principal Investigator proposes to perform a pilot study assessing the benefit-risk ratio of Remimazolam (a novel benzodiazepine with a short half-life) in the critical care units of Nantes University Hospital during the COVID-19 pandemic.

DETAILED DESCRIPTION:
The worldwide COVID-19 pandemic has led to a dramatic increase in the number of patients hospitalized in intensive care units for an acute respiratory failure in all countries. This situation has quickly led to massive shortage in masks, mechanical ventilation machines and common medications such as hypnotics. The reasons for such shortage are multiple: dramatic increase of the demand, production discontinuation because of shutdowns in multiple countries, and withholding of products by producing countries. All countries over the world are currently experiencing a major shortage in basic hypnotic medications (propofol, midazolam) in the intensive care as well as in the operating theatre. Remimazolam is a novel benzodiazepine with a short half-life that has been administered in patients undergoing major surgery, as well as in the intensive care unit. The Principal Investigator proposes to perform a pilot study assessing the benefit-risk ratio of Remimazolam in the critical care units of Nantes University Hospital during the COVID-19 pandemic.

ELIGIBILITY:
Inclusion Criteria:

* Patients at least 18 years old
* Inclusion in the first 96 hours after ICU admission, after clinical stabilization according to the attending physician's discretion.
* Expected duration of general anaesthesia ≥ 24 hours

Exclusion Criteria:

* Patients more than 85 years-old
* Refusal to participate
* Severe patients with moribund state within the 24 hours after admission to the ICU
* Withdrawal of Life Sustaining Therapies within the 24 hours after admission to the ICU
* Any pregnant or breast-feeding patient,
* Patients with known anaphylactic reactions to benzodiazepines, flumazenil, or a medical condition such that these agents are contraindicated (according to local label)
* Patients with allergy/hypersensitivity to bovine lactose, dextran or any other excipient in the remimazolam product
* Presence of acute alcoholic or illicit drug intoxication or benzodiazepine intoxication
* Inclusion in another clinical (drug) trial
* Patient under guardianship or trusteeship
* Patient under judicial protection
* Severe hepatic impairment defined as a Child-Pugh score > 10.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2020-11-30 (Actual); Primary Completion 2020-12-02 (Actual); Study Completion 2021-10-22 (Actual)

PRIMARY OUTCOMES:
composite endpoint including a combination of cardio-vascular and sedation events, from baseline (before infusion) to 8 hours, after the beginning of Remimazolam infusion | 8 hours after the beginning of infusion.
  For Safety: Cardiovascular event: Hypotension will be defined as a Mean Arterial Pressure ≤65mmHg or an increase ≥50% of the dose of norepinephrine (if appropriate), sustained over one hour after the beginning of Remimazolam.
  For Efficacy: Sedation event: the investigator will check if Remimazolam provides an adequate level of sedation assessed with the Richmond Assessment Sedation Scale. The level of sedation will be set by the attending physician and is usually set at-1/0. The investigator will also monitor the need to use standard hypnotic drugs within this time frame as further medication (propofol, midazolam, dexmedetomidine) in case of Remimazolam inefficacy (Richmond Assessment Sedation Scale).

SECONDARY OUTCOMES:
Adverse Events (all grades), related to Remimazolam. | 5 days
  An exhaustive monitoring of Adverse Events will be performed from Day-0 (inclusion), Day-1 and Day-2 (during infusion), to Day-5 (3 days after discontinuation).
Heart rate | 3 days
  Hemodynamic stability follow-up of heart rate, from day1 to day3.
Arterial pressure | 3 days
  Hemodynamic stability follow-up with systolic, diastolic and mean arterial pressure from day1 to day3.
Dose of norepinephrine | 3 days
  Hemodynamic stability follow-up with the dose of norepinephrine from day1 to day3.
Electrocardiogram (ECG) | 3 days
  Hemodynamic stability follow-up with electrocardiogram from day1 to day3.
Sedation. | 3 days
  The level of sedation will be assessed with clinical scale (Richmond Assessment Sedation Scale, scores from -5:unarousable to+4 : Combative or Bispectral Index, index from 100 (awake subject) to 0 (very deep sleep) .From day1 to day3.
Other sedatives. | 3 days
  The use or switch to other sedatives (midazolam, dexmedetomidine, propofol) in case of remimazolam inefficacy, will be monitored, from day1 to day3.
Wake-up time. | 3 days
  In minutes, defined as Richmond Assessment Sedation Scale 4 of -1/0, only in non-neurologic patients and if general anesthesia is definitely stopped at the end of remimazolam infusion.
Pharmacokinetics of Remimazolam and its metabolites (CNS 7054): Maximum Plasma Concentration. | 3 days
  maximum plasma concentration of Remimazolam and its metabolites, measured during the infusion and at the end. 9 Pharmacokinetic blood samplings during the infusion, and at Day-3, after Remimazolam discontinuation. In total 9 (nine) blood samples of 2 ml will be collected during the 48-hour infusion and during elimination phase (up to 24 hours post Remimazolam infusion).
Pharmacodynamics Remimazolam and its metabolites (CNS 7054): steady state plasma levels and elimination. | 3 days
  measured during the infusion and at the end. 9 Pharmacodynamics blood samplings during the infusion, and at Day-3, after Remimazolam discontinuation. In total 9 (nine) blood samples of 2 ml will be collected during the 48-hour infusion and during elimination phase (up to 24 hours post Remimazolam infusion).
Laboratory parameters : blood gas | 4 days
  Routine laboratory tests for blood gas will be made within this time frame: from day0 to day3.
Laboratory parameters: haemoglobin | 4 days
  Routine laboratory tests for haemoglobin will be made within this time frame: from day0 to day3.
Laboratory parameters: platelet count | 4 days
  Routine laboratory tests for platelet count will be made within this time frame: from day0 to day3.
Laboratory parameters: white blood cell count | 4 days
  Routine laboratory tests for white blood cell count will be made within this time frame: from day0 to day3.
Laboratory parameters: ionogram | 4 days
  Routine laboratory tests for ionogram will be made within this time frame: from day0 to day3.
Laboratory parameters: creatinine | 4 days
  Routine laboratory tests for creatinine will be made within this time frame: from day0 to day3.
Laboratory parameters: bilirubin | 4 days
  Routine laboratory tests for bilirubin will be made within this time frame: from day0 to day3.
Laboratory parameters: albumin | 4 days
  Routine laboratory tests for albumin will be made within this time frame: from day0 to day3.
Laboratory parameters: liver enzymes | 4 days
  Routine laboratory tests for liver enzymes will be made within this time frame: from day0 to day3.
Laboratory parameters: phosphorus | 4 days
  Routine laboratory tests for phosphorus will be made within this time frame: from day0 to day3.
Laboratory parameters: magnesium | 4 days
  Routine laboratory tests for magnesium will be made within this time frame: from day0 to day3.
Extubation failure defined as the need to intubate a patient in the 96 hours following extubation. | 28 days
  Extubation failure will be defined as the need to intubate a patient in the 96 hours following extubation.
Length of Mechanical ventilation. | 28 days
  Defined as the duration between the initiation and the successful weaning of mechanical ventilation. From Day-1 to ICU discharge or Day-28
Death. | 28 days
  in the ICU or at Day-28 if the patient is not discharged

CONTACTS AND LOCATIONS:
Overall Officials: Raphaël CINOTTI, MD, Principal Investigator — Nantes University Hospital
Locations (1):
- CHU de Nantes, Nantes, France

REFERENCES:
- [Derived] Grillot N, Vourc'h M, Hourmant Y, Bouras M, Rozec B, Rouhani A, Stoehr T, Jobert A, Roquilly A, Cinotti R. A phase 2 open-label pilot study of Remimazolam for sedation in critically ill patients. Anaesth Crit Care Pain Med. 2025 May;44(3):101510. doi: 10.1016/j.accpm.2025.101510. Epub 2025 Mar 31. PMID 40174701